CLINICAL TRIAL: NCT02184858
Title: Dose Titration Study to Test Efficacy and Safety of Lisinopril in Children Aged 1 to 18 Years With Primary or Secondary Hypertension.
Brief Title: Dose Titration of Lisinopril in Children Aged 1 to 18 Years With Primary or Secondary Hypertension
Acronym: Lisi-ped
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC project number: 2012/498; 2012-002927-14 (EudraCT Number)
Record Dates: First submitted 2014-06-10; First posted 2014-07-09 (Estimated); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Primary Hypertension; Secondary Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — Lisinopril; Angiotensin-Converting Enzyme Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- lisinopril (Experimental): dose titration of investigational product (lisinopril) dependant on blood pressure, levels of renin and aldosterone and on adverse events.
  Interventions: Drug: lisinopril, ACE-inhibitor

INTERVENTIONS:
Drug: lisinopril, ACE-inhibitor — Lisinopril 0.1mg/kg/d, titration with + 0.1mg/kg/d. Max; daily dose: 0.4mg/kg. CAVE: dose reduction in case of renal impairment

SUMMARY:
This open label 4 month study will evaluate efficacy (blood pressure lowering effects) and safety of lisinopril in children 1-18y whose parents grant permission to participate. This dose titration study is being conducted to support the statement that personalized titration of lisinopril (based on blood pressure and renin-aldosterone ratio) can increase patient response.

ELIGIBILITY:
Inclusion Criteria:

* Parental consent must be granted
* Patient age: 1y - 18 y
* Documented diagnosis of hypertension as defined in the National Heart, Lung and Blood Institute (NHBLI) 4th report, 2004
* No reversible cause found on diagnostic work-up for hypertension
* Children older than 6y: 24h blood pressure monitoring confirms the diagnosis of hypertension

Exclusion Criteria:

* Pregnancy
* Sexually active girls can only be included in the trial if they use an adequate form of birth control; during and until 30 days after ending the trial
* Following abnormal laboratory values: Hyperkaliemia (serum potassium > 5.3mmol/L); Anemia (hemoglobin < 8g/dL); AST or ALT > 3 times the upper limit of reference range; Total bilirubin > 3 times the upper limit of reference range
* Abnormalities of the oral cavity that can influence intake of medication
* Known sensitivity to ACE-inhibitors
* Known lactose intolerance
* History of angioedema
* Unilateral or bilateral stenosis of the renal artery
* Diagnosis of heart failure (NYHA Class II-IV)
* History of coarctation of the aorta
* Current treatment with: other drugs influencing the renin-angiotensin-aldosterone system; lithium; potassium sparing diuretics; non-steroidal anti-inflammatory drugs; aspirin; oral antidiabetic medication

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2014-06-25 (Actual); Primary Completion 2017-05-08 (Actual); Study Completion 2018-09-17 (Actual)

PRIMARY OUTCOMES:
blood pressure | 4 months

SECONDARY OUTCOMES:
Serum concentrations will be assessed after every dose titration | trough and 4 hours post dosing
Adverse events with assessment of specific blood parameters | up to 4 months
  sodium, potassium, creatinine, bilirubin, aspartate transaminase/alanine transaminase (AST/ALT) and blood count

CONTACTS AND LOCATIONS:
Overall Officials: Johan Vande Walle, PhD MD, Principal Investigator — Ghent University, Department of Pediatrics and Medical Genetics
Locations (1):
- Department of Pediatrics and Medical Genetics, Ghent, Belgium

REFERENCES:
- [Derived] Sandra L, Degraeuwe E, De Bruyne P, De Baere S, Croubels S, Van Bocxlaer JFP, Raes A, Vande Walle J, Gasthuys E, Vermeulen A. Population pharmacokinetics of lisinopril in hypertensive children and adolescents with normal to mildly reduced kidney function. Br J Clin Pharmacol. 2024 Feb;90(2):504-515. doi: 10.1111/bcp.15936. Epub 2023 Nov 10. PMID 37864281